CLINICAL TRIAL: NCT03430596
Title: a Pilot Study of Pramipexole to Treat Extrapyramidal Symptoms Induced by Antipsychotics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Wenjuan YU, director, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17411970300
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Extrapyramidal Syndrome
Keywords: Extrapyramidal syndromes praminpexole pilot study
MeSH Terms: conditions — Basal Ganglia Diseases | interventions — Pramipexole; Trihexyphenidyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- pramipexole (Experimental): pramipexole ,flexible dose (0.375mg/d-0.75mg/d)
  Interventions: Drug: Pramipexole
- Antan (Active Comparator): Antan,flexible dose (2-4mg/d)
  Interventions: Drug: Trihexyphenidyl hydrochloride

INTERVENTIONS:
Drug: Pramipexole — The dose of pramipexole range from 0.375mg/d to 0.75mg/d , The accurate dose of pramipexole can be adjusted by the patient's condition and tolerance .
  Other Names: SenForro
  Arms: pramipexole
Drug: Trihexyphenidyl hydrochloride — he dose of Antan range from 2 mg/d to 4 mg/d , The accurate dose of pramipexole can be adjusted by the patient's condition and tolerance .
  Other Names: Antan
  Arms: Antan

SUMMARY:
This study is a pilot phased interventional clinical trial . The first stage will recruit 10 patients with antipsychotic induced extrapyramidal symptoms.The patients will take pramipexole for 8 weeks. The inital dose of pramipexole will be 0.375 mg/d, and the adjustment of drug dose will be depended on the the doctor's decision and patients' condition.

The second stage was a randomized, rater blindness and Antan controlled clinical study. Researchers will recruit another 40 patients with extrapyramidal symptoms (tradive dyskinesia will be excluded). The patients will randomly be divided into artane group or pramipexole group, and the efficacy and safety condition of pramipexole and artane for different kinds of EPS will be compared. The pramipexole group will have 20 cases, and 20 cases of artane group. The dose of pramipexole group group range from 0.375mg/d to 0.75mg/d dose .The dose of artane range from 2 mg/d to 4 mg/d,.The accurate drug doses can be adjusted by the doctor according to the patients' condition .

Researchers will evualate patients' symptom at baseline, after three days' of baseline, 2 weeks,4 weeks, 6 weeks and 8 weeks. The Simpson-Angus Scale(SAS) 、Barnes Akathisia Rating Scale（BARS）,Abnormal Involuntary Movement Scale (AIMS), Positive and Negative Syndrome Scale(PANSS), Calgary Depression Scale for Schizophrenia(CDSS), Clinical Global Impression-severity of Illness Scale(CGI-S) will be evualated by the trained raters indicated as the drug's efficacy of the extrapyramidal symptoms and schizophrenia .The adverse events, laboratory parameters, vital signs, ECG will be recorded as the safety indicators of the study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-65 years old, male or female
2. Subjects who met DSM-IV-TR criteria for extrapyramidal symptoms
3. Scored 1 (mild) on at least two SAS items or 2 (moderate) on one of the items Exclusion Criteria are considered as antipsychotic induced parkinson ; Scored at least 2 (mild) on the BARS global item are considered as antipsychotic induced akathisia
4. Written informed consent provided by legal guardians or patients
5. Understand and voluntarily participate in this trail

Exclusion Criteria:

1 A history of severe nervous system disease or nervous system injury 2 A history of severe or unstable heart, liver, kidney, endocrine (including thyroid function), hematological (such as those with hemorrhagic tendency) condition 3 Subjects who have an imminent risk of suicideor who can be a threat to himself others which judged by investigator 4 Substance or alcohol dependence at enrolment 5 Pregnancy or lactation or willing to pregnant during the trial 6 Low compliance to the doctor 7 Subjects who can't take drug in time according to doctors' advice 8 scored (mild) on at least two AIMS items or 3 (moderate) on one of the items are considered as tardive dyskesia Withdrawl Criteria

1. An adverse sffecr or serious adverse effect occured so that the intervention needs to be stopped
2. Subjects with poor compliance or who didn't take drugs for 4 days
3. Obvious plan violation ,or the safety codition and symptoms of the patients are deteriorating
4. scored (mild) on at least two AIMS items or 3 (moderate) on one of the items are considered as tardive dyskesia
5. Researcher's decision of the withdrawl of the subjects -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The change of SAS BARS AIMS from baseline | 8 weeks
  To compare the condition of the extrapyramidal symptoms between two groups

SECONDARY OUTCOMES:
The change of PANSS CDSS CGI-S from baseline | 8 weeks
  To compare the change of the symptoms of chziophrenia between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, MD,Phd, Principal Investigator — Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Kelleher JP, Centorrino F, Huxley NA, Bates JA, Drake JK, Egli S, Baldessarini RJ. Pilot randomized, controlled trial of pramipexole to augment antipsychotic treatment. Eur Neuropsychopharmacol. 2012 Jun;22(6):415-8. doi: 10.1016/j.euroneuro.2011.10.002. Epub 2011 Dec 7. PMID 22153972
- [Background] Kasper S, Barnas C, Heiden A, Volz HP, Laakmann G, Zeit H, Pfolz H. Pramipexole as adjunct to haloperidol in schizophrenia. Safety and efficacy. Eur Neuropsychopharmacol. 1997 Feb;7(1):65-70. doi: 10.1016/s0924-977x(96)00393-8. PMID 9088887
- [Background] Ferger B, Buck K, Shimasaki M, Koros E, Voehringer P, Buerger E. Continuous dopaminergic stimulation by pramipexole is effective to treat early morning akinesia in animal models of Parkinson's disease: A pharmacokinetic-pharmacodynamic study using in vivo microdialysis in rats. Synapse. 2010 Jul;64(7):533-41. doi: 10.1002/syn.20759. PMID 20196139
- [Background] Kosmowska B, Wardas J, Glowacka U, Ananthan S, Ossowska K. Pramipexole at a Low Dose Induces Beneficial Effect in the Harmaline-induced Model of Essential Tremor in Rats. CNS Neurosci Ther. 2016 Jan;22(1):53-62. doi: 10.1111/cns.12467. Epub 2015 Oct 13. PMID 26459182
- [Background] Lorenc-Koci E, Wolfarth S. Efficacy of pramipexole, a new dopamine receptor agonist, to relieve the parkinsonian-like muscle rigidity in rats. Eur J Pharmacol. 1999 Nov 26;385(1):39-46. doi: 10.1016/s0014-2999(99)00704-9. PMID 10594343